CLINICAL TRIAL: NCT01712633
Title: Imaging Techniques in fMRI and fMRI Reproducibility: An NIH/FDA Interagency Collaboration
Brief Title: Tests of Functional Magnetic Resonance Imaging Techniques
Status: Terminated | Type: Observational
Why Stopped: Changes to funding
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 130003; 13-CC-0003
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Healthly Volunteers
Keywords: fMRI; Brain Perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Volunteers: Healthy Volunteers

SUMMARY:
Background:

- Functional magnetic resonance imaging (fMRI) is used to study the brain. It takes a series of pictures that can be used to look at how the brain processes information. It is used to study problems with thinking, language, and movement, among other things. Researchers are working to develop new and better fMRI techniques. To test these techniques, they want to perform fMRI scans on healthy volunteers.

Objectives:

- To test different fMRI techniques in healthy volunteers.

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will have fMRI scans of the brain. During these scans, they will be asked to perform simple tasks. These tasks may involve language, thinking, or motor skills. The scanning sessions will last up to 2 hours.
* Participants may be asked to return for additional fMRI scans over several years.

DETAILED DESCRIPTION:
Functional magnetic resonance imaging (fMRI) is a non invasive imaging technique that enables scientists to understand the biological basis of higher order cognitive functioning such as emotions, attention, language and visual processing. It has been used as a research tool since the 1980 s. Recently, fMRI has received approval by the Center for Medicare and Medicaid Services (CMS) to be used clinically which we believe will drastically increase its use in clinical decision making by physicians in the very near future. However, currently implemented imaging techniques have technical and physiologic limitations such as susceptibility artifacts, image distortions, physiological noise, and MRI induced energy deposition from radiomagnetic waves typically used in fMRI acquisitions that may potentially reduce the clinical effectiveness of this imaging modality. This protocol is a unique technical development pilot study being conducted jointly by researchers at the National Institutes of Health (NIH) and the US Food and Drug Administration (FDA) to evaluate the performance of physiologic and technical factors of fMRI imaging methods and equipment that may affect image quality, reproducibility, and reliability in the clinical setting. These studies are an important basis upon which improved regulatory evaluation of new functional imaging technologies can be performed as these technologies become increasingly used in patient care in the future.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy volunteers, new or from current NIH protocols are eligible. Healthy volunteers will be defined according the history obtained from reported medical history, medical record (reported at registration), the MRI safety questionnaire, and a clinical grade noncontrast brain MRI.
* Willing to travel to the NIH for follow-up visits
* Greater than 18 years old
* Able to understand and sign informed consent.
* Bilingual or multilingual subjects can participate in this study as long as the subjects are also fluent in English. Subjects do not need to be native or monolingual speakers of English.

EXCLUSION CRITERIA:

The following criteria will be used to exclude subjects from participating in this protocol:

* Implanted metal clips or wires of the type which may concentrate radiofrequency fields or cause tissue damages from twisting in a Magnetic field. Examples:

  * Aneurysm clip, implanted neural stimulator,
  * Implanted cardiac pacemaker, defibrillator, or certain other implanted electrical or metallic devices,
  * Cochlear implant, ocular foreign body (metal shavings),
  * Any implanted device (pumps, infusion devices, etc.),
  * Shrapnel injuries,
  * History of metal in head or eyes or other parts of the body.
  * Vagus Nerve Stimulators (VNS)
  * Subjects with tattoos that contain metal.
* Pregnant women
* Over 350 lbs because of the weight limit of the MRI table
* Prior surgery that may render performing the MRI to be unsafe.
* Untreatable claustrophobia otherwise requiring anesthesia or antianxiety medications that may alter the subject s ability to perform the tasks during fMRI scanning.
* Subjects will be asked to refrain from drinking or eating caffeinated foods or drinks the morning of the scan that can result in vessel vasoconstriction prior to the scan.
* Any contraindications that the Physician identifies from the Subject s reported history, MRI Safety Questionnaire and/or medical record.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers willing to come to NIH or are already part of an existing NIH protocol.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
evaluation of fMRI techniques | Study day 1, followup visit(s)
  To test different fMRI techniques in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia M Biassou, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hennig J, Speck O, Koch MA, Weiller C. Functional magnetic resonance imaging: a review of methodological aspects and clinical applications. J Magn Reson Imaging. 2003 Jul;18(1):1-15. doi: 10.1002/jmri.10330. PMID 12815634
- [Background] Bennett CM, Miller MB. How reliable are the results from functional magnetic resonance imaging? Ann N Y Acad Sci. 2010 Mar;1191:133-55. doi: 10.1111/j.1749-6632.2010.05446.x. PMID 20392279
- [Background] Pillai JJ. The evolution of clinical functional imaging during the past 2 decades and its current impact on neurosurgical planning. AJNR Am J Neuroradiol. 2010 Feb;31(2):219-25. doi: 10.3174/ajnr.A1845. PMID 20150316
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-CC-0003.html